CLINICAL TRIAL: NCT04218591
Title: A Study on the Effect of Platelet Rich Plasma (PRP) on Osteoarthritis in the Thumb Base
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Maria Wilcke, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP vs placebo
Record Dates: First submitted 2019-12-19; First posted 2020-01-06 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Thumb Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP (Active Comparator): Intra-articular injection PRP
  Interventions: Other: PRP
- Saline (Placebo Comparator): Intra-articular injection Saline
  Interventions: Other: Placebo

INTERVENTIONS:
Other: PRP — Platelet rich plasma
  Arms: PRP
Other: Placebo — Saline
  Arms: Saline

SUMMARY:
Randomized comparison between Platelet Rich Plasma (PRP) and placebo (Saline) for thumb base.osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Arthritis in the thumb base.
* Radiological Eaton Littler class 1-3.
* Clinical signs of thumb base osteoarthritis: pain at palpation of the CMC-1 joint and pain during provocation/grinding test.

Exclusion Criteria:

* Rheumatoid arthritis.
* Ongoing infection in the hand or wrist.
* History of gout or pseudo gout.
* Inability to co-operate with the follow-up protocol (language difficulties, severe psychiatric disorder, cognitive impairment, drug addiction).
* Intra-articular injection in the affected joint within 6 months.
* Eaton Littler class 4 (STT joint involved).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in patient-rated pain on load | 3 and 6 months after injection.
  Numerical rating scale 0-10p (10=worst possible pain).

SECONDARY OUTCOMES:
Change in Nelson Thumb score | 3 and 6 months after injection.
  Patient Rated Outcome Measure, 0-100p, lower score= more disability
Change in EQ-5D | 3 and 6 months after injection.
  Weight mean value: 0=dead, 1= healthy
Change in Patient-rated Wrist and Hand Evaluation (PRWHE) | 3 and 6 months after injection.
  Patient Rated Outcome Measure 0-100p, higher score=more disability
Change in Disability of the Hand, Arm and Shoulder (DASH) score | 3 and 6 months after injection.
  Patient Rated Outcome Measure, 0-100p higher score=more disability
Change in Hospital Anxiety and Depression Score (HADS), | 3 and 6 months after injection.
  2 subscores for anxiety (0-21p) and depression (0-21p), higher score = worse
Change in Pain Catastrophizing Score (PCS). | 3 and 6 months after injection.
  0-52p, higher score = more pain catastrophizing
Change in thumb range of motion | 3 and 6 months after injection.
  Radial and palmar abduction of the first metacarpal (degrees)
Change in thumb strength | 3 and 6 months after injection.
  Key pinch and pinch strength (Kg)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Wilcke, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Hand Surgery Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No